CLINICAL TRIAL: NCT00435565
Title: Severe Hypoglycemia in Pregnant Women With Type 1 Diabetes. Incidence, Risk Markers and Possibilities for Prevention
Brief Title: Severe Hypoglycemia in Pregnant Women With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Other Study IDs: ringholm
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2007-02-15 (Estimated); Status verified 2007-02

CONDITIONS: Pregnancy; Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Background:

The risk of stillbirth and preterm delivery is three times increased among pregnant women with type 1 diabetes compared with healthy pregnant women. Normal blood glucose levels are mandatory in order to prevent these complications. Severe hypoglycemia (requiring assistance from another person) is the decisive limiting factor for obtaining near-normal blood glucose regulation in pregnant women with type 1 diabetes. Severe hypoglycemia occurs in about one third of pregnancies complicated with type 1 diabetes and can result in unconsciousness, traffic accidents and deaths.

Aim: To test the following hypotheses:

1. Severe hypoglycemia is frequent in pregnancy complicated by type 1 diabetes with the highest incidence in gestational weeks 8-16 and the lowest incidence in gestational weeks 28-34
2. Predictors for severe hypoglycemia during pregnancy complicated with type 1 diabetes can be identified at the first pregnancy visit
3. Possible pathophysiological mechanisms include changes in the growth hormone system and in the renin-angiotensin-system during pregnancy

Methodology:

One hundred and eight pregnant women with type 1 diabetes are consecutively and prospectively included. In connection with the clinical control at the first pregnancy visit at week 9 and in gestational weeks 14, 22, 28, 34 and one day postpartum the following tests are carried out:

The patients are asked to answer a validated questionnaire about mild and severe hypoglycemia and hypoglycemia-associated factors such as blood glucose level during hypoglycemia, the degree of awareness, pregnancy-associated nausea and vomiting, insulin type and dose etc. Other medication, exercise habits, coffee- and alcohol intake, smoking and social status will be recorded. In case of severe hypoglycemia a structured interview concerning the episode will be performed within 24 hours. Blood glucose, HbA1c, the degree of insulin resistance and the levels of IGF1, placenta growth hormone and of the renin-angiotensin-system will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Pregnancy before gestational week 14

Exclusion Criteria:

* Other diseases that might influence the risk of severe hypoglycemia

Sex: Female
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Lene R Nielsen, MD, Principal Investigator — Rigshospitalet, Denmark